CLINICAL TRIAL: NCT06960460
Title: Prospective, Multicenter, European Clinical Investigation Evaluating the Short and Medium-term Performance and Safety of the Global D ZygoFixU Implant-prosthetic System
Brief Title: Study Evaluating the Performance and Safety in the Medium and Long Term of Global D ZygoFixU System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2302-G-ZYGO-C
Record Dates: First submitted 2025-04-02; First posted 2025-05-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Dental Implants
Keywords: dental implant; survival rate; zygomatic; performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZygoFixU system (Experimental): Adult male or female patient, requiring implant treatment with Global D zygomatic implants (placement of two or four implants),
  Interventions: Other: Dental implant surgery with ZygoFixU implants

INTERVENTIONS:
Other: Dental implant surgery with ZygoFixU implants — Adult patients who have had dental implant surgery.

SUMMARY:
Global D has developed an zygomatic implant prosthetic system (ZygoFixU range): zygomatic implants, prosthetic parts and associated instruments. These devices have a design similar to other zygomatic implants on the market and are therefore not innovative. These non-CE marked devices are assessed during investigation 2302-G-ZYGO-C for their performance and for their short- and medium-term safety. These implants will be placed using specific instruments, by oral or cranio-maxillofacial surgeons with significant experience in the placement of zygomatic implants and trained in clinical research.

DETAILED DESCRIPTION:
Study design: Interventional pivotal study involving humans, prospective with continuous series, multicentre, European, open-label, non-comparative.

Clinical investigation classification: class 2 clinical investigation according to ANSM in France, aiming at establishing the conformity of a class IIb, non CE-marked medical device. Clinical investigation to demonstrate device compliance, in accordance with Article 62.1 of the MDR.

Investigators: Patient recruitment and follow-up will be carried out by dental surgeons or oral surgeons/stomatologists in France and Italy. 11 sites will participate in the CI in 2 countries (Italy and France).

Objective: To assess the performance of the ZygoFixU implant-prosthetic system by measuring the survival rate at 1 year postoperatively.

Population: Adult male or female patients, whose growth and development of the maxillary bone is complete, partially or completely edentulous with advanced atrophy of the maxillary bone (grades IV, V and VI according to the Cawood and Howell classification if used).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient,
* Patient whose growth and development of the maxillary bone is complete according to the investigator's judgement,
* Partially or completely edentulous patient,
* Patient with advanced maxillary atrophy (grades IV, V and VI according to the Cawood and Howell classification if used),
* Patient requiring implant treatment with Global D zygomatic implants (placement of two or four implants),
* Patient with acceptable oral opening (>3 cm measured anteriorly),
* Patient able to read, understand and answer the quality-of-life questionnaire of the investigation and able to give consent,
* Patient agreeing to comply with the protocol design and to send his/her follow-up data, even in the event of a move,
* Patient having signed the consent form,
* In France, patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient's state of health at enrolment:

  * General contraindications to implant surgery
  * Patient with zygomatic bone disease
  * Patient with untreated periodontal disease
  * Patient with acute or chronic infection in the implant placement area, or systemic infection, including acute or chronic maxillary sinusitis
  * Patient with acute or chronic inflammation in the implant placement area, or systemic inflammation,
  * Patient with uncontrolled diabetes (unstable blood glucose)
  * Patient with immunodeficiencies or using immunosuppressants
  * Patient who received radiation of more than +70 Gy to the head and neck region
  * Patient using intravenous aminobisphosphonates within 5 years prior to surgery
* Patient who are smokers (>10 cigarettes/day) or with alcohol or drug addiction
* Person placed under legal protection (this includes guardianship, curatorship and legal protection).
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the performance of the ZygoFixU implant-prosthetic system by measuring the survival rate at 1 year postoperatively. | 1 year
  Measurement of the survival rate of Global D zygomatic implants 1 year after the surgical procedure by the rate of in situ implants.

SECONDARY OUTCOMES:
To assess the performance of the ZygoFixU implant-prosthetic system via the survival rate | 2, 3, 4 years and 5 years
  Measurement of performance by the survival rate of Global D zygomatic implants at 2, 3, 4 years and 5 years postoperatively
the success rate at 1 year postoperatively, 2, 3, 4 years and 5 years postoperatively - the quality of life of patients preoperatively, at 6-8 months postoperatively, 1 year postoperatively, 2, 3, 4 years and 5 years postoperatively. | 12 months, 2, 3, 4 years and 5 years
  The success rates at 12 months, 2, 3, 4 years and 5 years respectively defined by complication and failure indicators (implant mobility, continuous radiolucency around the implant, peri-implantitis with/without suppuration leading to implant failure, fracture of the implant or prosthetic components, pain, dysaesthesia, foreign body sensation, persistent oedema (periorbital region), persistent maxillary sinus infection leading to implant failure, postoperative hematoma, postoperative infection, postoperative suppuration)
To assess the safety of the ZygoFixU implant-prosthetic system via: - immediate and delayed complications (adverse device events and effects, defects) | 2, 3, 4 years and 5 years
  The survival rate at 2, 3, 4 years and 5 years postoperatively - The number and rate of serious and non-serious biological and technical complications reported as related to the use of Global D zygomatic implants and/or prosthetic parts throughout patient follow-up
To assess surgeon satisfaction with the use of the ZygoFixU implant-prosthetic system. | After surgery
  Measurement of surgeon satisfaction with all devices used by an investigation-specific questionnaire (without score scale), completed after surgery.
To assess patient satisfaction with the ZygoFixU implant-prosthetic system | 1 year
  Measurement of patient satisfaction by an investigation-specific questionnaire completed 12 months postoperatively (without score scale).
To assess the safety of the ZygoFixU implant-prosthetic system via: - immediate and delayed complications (adverse device events and effects, defects) | 2, 3, 4 years and 5 years
  Manual stability at all patient follow-up visits: the practitioner exerts slight pressure to check that the implant-prosthetic system does not move. A stable implant is an immobile implant

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - CCOI Toulouse, Toulouse, France
  - Cabinet dentaire Dr HADJ, Marseille
- Université de Bologne, Bologne, Italie, Italy

IPD SHARING:
Plan to Share IPD: No